CLINICAL TRIAL: NCT02309099
Title: Cochlear Implantation After Labyrinthectomy or a Translabyrinthine Surgical Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Med-El Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-1818
Record Dates: First submitted 2014-11-12; First posted 2014-12-05 (Estimated); Results first posted 2018-12-10 (Actual); Last update posted 2019-01-07 (Actual); Status verified 2018-01

CONDITIONS: Unilateral Acoustic Neuroma; Meniere's Disease
Keywords: Acoustic Neuroma; Vestibular Schwannoma; Meniere's Disease
MeSH Terms: conditions — Neuroma, Acoustic; Meniere Disease | interventions — Cochlear Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cochlear Implant (Experimental): Cochlear implantation of the affected ear
  Interventions: Device: Cochlear Implant

INTERVENTIONS:
Device: Cochlear Implant — Cochlear implantation used a treatment for single-sided deafness resultant of labyrinthectomy or a translabyrinthine surgical approach
  Other Names: MED-EL CONCERT cochlear implant system; MED-EL SYNCHRONY cochlear implant system

SUMMARY:
The goal of this project is to determine whether subjects who have undergone labyrinthectomy or a translabyrinthine surgical approach as the treatment for vestibular schwannoma or Meniere's disease benefit from cochlear implantation on speech perception and localization tasks.

If the auditory nerve is able to transmit this signal effectively, then these two populations may be able to utilize the combination of electric (in the affected ear) and acoustic (in the non-affected ear) information for improved speech perception in noise and localization as reportedly experienced in other unilateral sensorineural hearing loss populations.

DETAILED DESCRIPTION:
The treatment for cases of vestibular schwannoma or Meniere's disease may require a translabyrinthine surgical approach. This surgical approach results in a complete loss of hearing in the surgical ear, leaving the patient with a unilateral hearing loss. Though assistive hearing technologies exist to route signals from the poorer hearing ear to the better hearing ear, affected patients continue to have limitations with localization and speech perception in noise. An alternative hearing device is a cochlear implant, which would provide the signal to the affected ear. This could potentially offer binaural cues, thus improving localization and speech perception in noise. Since the surgical procedures for a translabyrinthine approach parallel those for cochlear implantation, insertion of the cochlear implant could occur within the same surgery.

A vestibular schwannoma is a benign tumor on cranial nerve VIII that affects the vestibular and auditory systems. Hearing loss on the side of the vestibular schwannoma may result from degeneration of hair cells and spiral ganglia or growth of the schwannoma into the cochlear space. Treatment options include observation from routine imaging, radiation therapy, or surgical removal of the tumor. Despite treatment for the vestibular schwannoma, auditory sensitivity may be further reduced on the affected side as a result of the radiation therapy or compromises to the inner ear or cranial nerve VIII from surgical removal. Thus, in cases of unilateral vestibular schwannoma the patient is often left with a unilateral profound hearing loss.

Patients who are scheduled to undergo labyrinthectomy for intractable Meniere's disease are a second population with resulting unilateral profound hearing loss. These patients typically have non-functional hearing on the affected ear prior to the procedure. The main indication for the surgery is intractable vertigo and thus the loss of already non-functional hearing is typically well accepted.

Though hearing on the contralateral ear may be within normal limits, unilateral hearing loss is known to result in reduced speech perception in noise, variable abilities on localization tasks, increased report of hearing handicap, and reduced quality of life. Due to the severity of the hearing loss, these patient populations cannot utilize conventional amplification that would offer auditory input to the affected ear. The current hearing device options for this patient population include contralateral routing of signal (CROS) hearing aids and bone-conduction devices. With a CROS hearing aid, a microphone positioned near the affected ear picks up the signal and sends it to a hearing aid placed on the contralateral ear to present the signal to the unaffected side. Bone-conduction devices transmit the signal from the affected ear to the contralateral ear via transcutaneous vibrations. Though CROS hearing aids and bone-conduction devices provide the patient with auditory information from both sides, the ability to use binaural cues for localization and speech perception in noise is variable.

It is of interest as to the potential benefit of cochlear implantation in these populations considering the profound hearing loss resulting from surgical intervention. A cochlear implant is a two-part system, including the internal electrode array and external speech processor. The internal electrode array is surgically implanted into the affected cochlea. The external speech processor receives sounds and transmits this signal to the internal portion. The electrode array presents the signal via electrical pulses within the cochlear space, which is interpreted by the brain as sound.

Cochlear implantation has been reported as a viable treatment option in other cases of unilateral hearing loss, including sudden sensorineural hearing loss, and severe tinnitus. Further, cochlear implantation has been shown to offer superior speech perception in noise, localization abilities, and subjective report in cases of unilateral sensorineural hearing loss as compared to CROS hearing aids and bone-conduction devices.

There is limited evidence as to the success of cochlear implantation in patients with unilateral profound hearing loss resulting from vestibular schwannoma. One study reported variable speech perception outcomes in five cochlear implant recipients with a history of vestibular schwannoma due to neurofibromatosis type 2 (NF2) or sporadic growth. Limitations of this study are the subjects underwent a range of treatments prior to cochlear implantation and the cases reviewed had profound hearing loss in both ears. A second study reported on a case study of unilateral vestibular schwannoma removal and simultaneous cochlear implantation. This subject reportedly experienced an improvement in speech perception abilities and quality of life postoperatively. Determining the preferred treatment option for patients suffering from unilateral vestibular schwannoma is still needed.

Further, there is limited evidence of the preferred treatment option for patients suffering from unilateral profound hearing loss after undergoing a labyrinthectomy for intractable Meniere's disease. One study reported on a patient who underwent bilateral labyrinthectomies for Meniere's disease. They reported an improvement in speech perception abilities and subjective benefit; however, there was a delay between the two surgeries. Allowing for a waiting period between the two surgeries is not ideal as cochlear ossification may occur, limiting the ability to successfully insert the electrode array. Another study also reported successful outcomes from cochlear implantation in subjects with bilateral Meniere's disease. However, there is no published report investigating whether cochlear implantation improves speech perception and/or localization abilities in unilateral cases of Meniere's disease.

The goal of this project is to determine whether subjects who have undergone labyrinthectomy or a translabyrinthine surgical approach as the treatment for vestibular schwannoma or Meniere's disease benefit from cochlear implantation on speech perception and localization tasks. If the auditory nerve is able to transmit this signal effectively, then these two populations may be able to utilize the combination of electric (in the affected ear) and acoustic (in the non-affected ear) information for improved speech perception in noise and localization as reportedly experienced in other unilateral sensorineural hearing loss populations.

ELIGIBILITY:
Inclusion Criteria:

1. Scheduled to undergo a surgical procedure that will result in profound hearing loss in the surgical ear [unilateral vestibular schwannoma wtih planned translabyrinthine surgery or unilateral Meniere's disease with planned labyrinthectomy] [diagnosed by UNC investigators]
2. Pure-tone average (PTA) less than or equal to 35 decibels Hearing Level (dB HL) in the contralateral ear [no evidence of retrocochlear dysfunction]
3. Unaided consonant-nucleus-consonant (CNC) words score greater than or equal to 80% in the contralateral ear
4. Greater than 18 years of age at implantation
5. Realistic expectations
6. Willing to obtain appropriate meningitis vaccinations
7. No reported cognitive issues [pass the Mini Mental State Examination screener]
8. Able and willing to comply with study requirements, including travel to investigational site
9. Obtain Centers for Disease Control and Prevention (CDC) recommended meningitis vaccinations prior to surgery

Exclusion Criteria:

1. History of implantable technology in either ear, such as a bone-conduction implant
2. Non-native English speaker [speech perception materials presented in English]
3. Inability to participate in follow-up procedures (unwillingness, geographic location)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2017-11-08 (Actual); Study Completion 2017-11-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Brown, MD, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Background] Lustig LR, Yeagle J, Niparko JK, Minor LB. Cochlear implantation in patients with bilateral Meniere's syndrome. Otol Neurotol. 2003 May;24(3):397-403. doi: 10.1097/00129492-200305000-00009. PMID 12806291
- [Background] Osborn HA, Yeung R, Lin VY. Delayed cochlear implantation after surgical labyrinthectomy. J Laryngol Otol. 2012 Jan;126(1):63-5. doi: 10.1017/S0022215111002374. Epub 2011 Sep 14. PMID 21914249
- [Background] Pai I, Dhar V, Kelleher C, Nunn T, Connor S, Jiang D, O'Connor AF. Cochlear implantation in patients with vestibular schwannoma: a single United Kingdom center experience. Laryngoscope. 2013 Aug;123(8):2019-23. doi: 10.1002/lary.24056. Epub 2013 Apr 24. PMID 23616085
- [Background] Wareing MJ, O'Connor AF. The role of labyrinthectomy and cochlear implantation in Meniere's disease. Ear Nose Throat J. 1997 Sep;76(9):664-6, 668, 671-2. No abstract available. PMID 9309909
- [Background] Zanetti D, Campovecchi CB, Pasini S, Nassif N. Simultaneous translabyrinthine removal of acoustic neuroma and cochlear implantation. Auris Nasus Larynx. 2008 Dec;35(4):562-8. doi: 10.1016/j.anl.2007.11.011. Epub 2008 Feb 19. PMID 18243617

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was completed in medical clinic by surgeon if a patient is identified as a potential participant and has decided to undergo vestibular schwannoma resection via a translabyrinthine surgical approach or a labyrinthectomy for Meniere's disease.
Pre-assignment Details: Groups were based on the participants' diagnosis (vestibular schwannoma or Meniere's disease) and subsequent surgery. Participants were initially consented into their specific group.
Groups:
- Vestibular Schwannoma: Diagnosis of vestibular schwannoma. Within the resection surgery via translabyrinthine surgical approach, cochlear implantation occurred following surgeon's visual confirmation of anatomically intact auditory nerve.
- Meniere's Disease: Diagnosis of Meniere's disease. During the labyrinthectomy surgery, cochlear implantation was completed following labyrinthectomy.
Period: Overall Study
Arm/Group | Vestibular Schwannoma | Meniere's Disease
Started | 7 | 3
Cochlear Implantation (Cochlear implantation following initial surgical procedure (schannoma resection or labyrinthectomy)) | 7 | 3
Initial Activation (Initial activation of cochlear implant (2-4 weeks following surgical procedure/implantation)) | 7 | 3
Cochlear Implant Use/Follow-Up (Device use over the initial 12 months following initial activation (1-month to 12-months)) | 5 (5 participants completed cochlear implant use/follow-up (2 did not complete due to adverse event)) | 3
Completed | 5 (5 participants completed the study (2 did not complete due to adverse event)) | 3
Not Completed | 2 | 0
Not completed — Adverse Event | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vestibular Schwannoma | Meniere's Disease | Total
Number analyzed (Participants) | 7 | 3 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 1 | 6
  >=65 years | 2 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 3 | 1 | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 3 | 10

OUTCOME MEASURES:

1. Primary Outcome: Change in Consonant-Nucleus-Consonant (CNC) Words Scores Over Time
Description: Testing open-set word understanding. Recorded CNC Words lists were presented to the participant while listening to the cochlear implant alone and contralateral ear plugged/masked. Resultant score is a percentage of words correct. A higher score is better.
Time Frame: Intervals within the first 12 months of device use
Population: Cochlear Implant Use/Follow-Up One participant in the Meniere's disease group did not complete the 12-month follow-up interval (protocol deviation) and is excluded from that analysis.
Measure: Mean (Full Range); unit: Percentage of words correct
Arm/Group | Vestibular Schwannoma | Meniere's Disease
Number analyzed (Participants) | 5 | 3
Percentage of words correct
  1-Month | 23.6 [0 to 72] | 22 [6 to 44]
  3-Month | 18.8 [2 to 46] | 42.7 [24 to 64]
  6-Month | 20.4 [4 to 34] | 48.7 [36 to 56]
  12-Month: number analyzed (Participants) | 5 | 2
  12-Month | 20.4 [0 to 52] | 45 [26 to 64]

2. Primary Outcome: Change in Arizona Biomedical Institute (AzBio) Sentences in Quiet Scores Over Time
Description: Testing open-set sentence understanding with no background noise present. Recorded AzBio Sentences lists were presented to the participant while listening with the cochlear implant on and contralateral ear open. Resultant score is a percentage of words correct. A higher score is better.
Time Frame: Intervals within the first 12 months of device use
Population: as for outcome 1
Measure: Mean (Full Range); unit: Percentage of words correct
Arm/Group | Vestibular Schwannoma | Meniere's Disease
Number analyzed (Participants) | 5 | 3
Percentage of words correct
  1-Month | 98.6 [97 to 100] | 99.7 [99 to 100]
  3-Month | 98.8 [96 to 100] | 99.3 [98 to 100]
  6-Month | 97.8 [96 to 99] | 99.7 [99 to 100]
  12-Month: number analyzed (Participants) | 5 | 2
  12-Month | 99.2 [98 to 100] | 99.5 [99 to 100]

3. Primary Outcome: Change in AzBio Sentences in Noise Scores (S0N0) Over Time
Description: Testing open-set sentence understanding with concurrent background noise present at 0 decibel signal-to-noise ratio (dB SNR). Recorded AzBio Sentences lists were presented to the participant while listening with the cochlear implant on and contralateral ear open; the speech and noise were colocated in this condition (S0N0). Resultant score is a percentage of words correct. A higher score is better.
Time Frame: Intervals within the first 12 months of device use
Population: as for outcome 1
Measure: Mean (Full Range); unit: Percentage of words correct
Arm/Group | Vestibular Schwannoma | Meniere's Disease
Number analyzed (Participants) | 5 | 3
Percentage of words correct
  1-Month | 33.2 [21 to 45] | 44 [28 to 54]
  3-Month | 29.4 [15 to 52] | 41.3 [24 to 55]
  6-Month | 30.2 [19 to 51] | 40.3 [26 to 54]
  12-Month: number analyzed (Participants) | 5 | 2
  12-Month | 42.2 [25 to 59] | 50.5 [47 to 54]

4. Primary Outcome: Change in AzBio Sentences in Noise Scores (S0NCI) Over Time
Description: Testing open-set sentence understanding with concurrent background noise present at 0 dB SNR. Recorded AzBio Sentences lists were presented to the participant while listening with the cochlear implant on and contralateral ear open; the speech was presented at 0 degrees azimuth and noise to the implanted side in this condition (S0NCI). Resultant score is a percentage of words correct. A higher score is better.
Time Frame: Intervals within the first 12 months of device use
Population: as for outcome 1
Measure: Mean (Full Range); unit: Percentage of words correct
Arm/Group | Vestibular Schwannoma | Meniere's Disease
Number analyzed (Participants) | 5 | 3
Percentage of words correct
  1-Month | 76.6 [67 to 88] | 84.7 [77 to 97]
  3-Month | 66.6 [37 to 88] | 85 [76 to 94]
  6-Month | 73.4 [49 to 94] | 83.3 [70 to 96]
  12-Month: number analyzed (Participants) | 5 | 2
  12-Month | 71.8 [53 to 90] | 82.5 [70 to 95]

5. Primary Outcome: Change in AzBio Sentences in Noise Scores (S0NContra) Over Time
Description: Testing open-set sentence understanding with concurrent background noise present at 0 dB SNR. Recorded AzBio Sentences lists were presented to the participant while listening with the cochlear implant on and contralateral ear open; the speech was presented at 0 degrees azimuth and noise to the contralateral ear in this condition (S0NContra). Resultant score is a percentage of words correct. A higher score is better.
Time Frame: Intervals within the first 12 months of device use
Population: as for outcome 1
Measure: Mean (Full Range); unit: Percentage of words correct
Arm/Group | Vestibular Schwannoma | Meniere's Disease
Number analyzed (Participants) | 5 | 3
Percentage of words correct
  1-Month | 21.6 [4 to 49] | 28 [16 to 51]
  3-Month | 12 [4 to 24] | 38 [17 to 50]
  6-Month | 18 [11 to 37] | 45 [17 to 60]
  12-Month: number analyzed (Participants) | 5 | 2
  12-Month | 25.4 [14 to 38] | 49 [42 to 56]

6. Primary Outcome: Change in Bamford-Kowal-Bench-Speech-in-Noise (BKB-SIN) Scores (S0N0) Over Time
Description: Testing open-set sentence understanding with concurrent background noise present at various levels. Recorded BKB-SIN lists were presented to the participant while listening with the cochlear implant on and contralateral ear open; the speech and noise were colocated in this condition (S0N0). Resultant score is the signal-to-noise ratio in decibels (dB SNR) at which the participant scores 50% of the target words correct. A lower score is better.
Time Frame: Intervals within the first 12 months of device use
Population: as for outcome 1
Measure: Mean (Full Range); unit: dB SNR
Arm/Group | Vestibular Schwannoma | Meniere's Disease
Number analyzed (Participants) | 5 | 3
dB SNR
  1-Month | -1.3 [-3 to 0.5] | -1 [-2 to 0.5]
  3-Month | -0.9 [-2.5 to 1] | -0.5 [-1 to 0]
  6-Month | 0.9 [-1 to 2.5] | -1.83 [-2 to -1.5]
  12-Month: number analyzed (Participants) | 5 | 2
  12-Month | -0.9 [-3 to 1] | -2 [-2 to -2]

7. Primary Outcome: Change in BKB-SIN Scores (S0NCI) Over Time
Description: Testing open-set sentence understanding with concurrent background noise present at various levels. Recorded BKB-SIN lists were presented to the participant while listening with the cochlear implant on and contralateral ear open; the speech was presented at 0 degrees azimuth and noise to the implanted side in this condition (S0NCI). Resultant score is the signal-to-noise ratio at which the participant scores 50% of the target words correct. A lower score is better.
Time Frame: Intervals within the first 12 months of device use
Population: as for outcome 1
Measure: Mean (Full Range); unit: dB SNR
Arm/Group | Vestibular Schwannoma | Meniere's Disease
Number analyzed (Participants) | 5 | 3
dB SNR
  1-Month | -3.5 [-5 to -1] | -6 [-7 to -5.5]
  3-Month | -3.4 [-6 to -0.5] | -5.2 [-6.5 to -4.5]
  6-Month | -3.3 [-6.5 to -1] | -5.33 [-5.5 to -5]
  12-Month: number analyzed (Participants) | 5 | 2
  12-Month | -4.4 [-7 to -2] | -5 [-6 to -4]

8. Primary Outcome: Change in BKB-SIN Scores (S0NContra) Over Time
Description: Testing open-set sentence understanding with concurrent background noise present at various levels. Recorded BKB-SIN lists were presented to the participant while listening with the cochlear implant on and contralateral ear open; the speech was presented at 0 degrees azimuth and noise to the contralateral ear in this condition (S0NContra). Resultant score is the signal-to-noise ratio at which the participant scores 50% of the target words correct. A lower score is better.
Time Frame: Intervals within the first 12 months of device use
Population: as for outcome 1
Measure: Mean (Full Range); unit: dB SNR
Arm/Group | Vestibular Schwannoma | Meniere's Disease
Number analyzed (Participants) | 5 | 3
dB SNR
  1-Month | 1.7 [1 to 3] | -1 [-2 to 0.5]
  3-Month | 1.8 [1 to 3] | -2.3 [-4 to 0]
  6-Month | 2.2 [1 to 3.5] | -1.3 [-2.5 to 0.5]
  12-Month: number analyzed (Participants) | 5 | 2
  12-Month | 1.2 [-0.5 to 2.5] | -0.25 [-1.5 to 1]

9. Primary Outcome: Change in Localization Root-mean-squared (RMS) Error Over Time
Description: Participants identified a speech-shaped noise source presented at various presentation levels within an 11-speaker array. Participants localized the sound source with the cochlear implant on and contralateral ear open. The RMS error (degrees) was estimated; a lower degree is more accurate/better localization of the sound source.
Time Frame: Intervals within the first 12 months of device use
Population: as for outcome 1
Measure: Mean (Full Range); unit: Degrees
Arm/Group | Vestibular Schwannoma | Meniere's Disease
Number analyzed (Participants) | 5 | 3
Degrees
  1-Month | 40.5 [30.3 to 51.2] | 30.7 [27 to 32.9]
  3-Month | 40.2 [27.4 to 51.4] | 25.7 [23.4 to 27]
  6-Month | 37.5 [26.2 to 55] | 21.5 [18.7 to 23.1]
  12-Month: number analyzed (Participants) | 5 | 2
  12-Month | 36.7 [18.5 to 54.5] | 20.3 [18.6 to 22]

10. Primary Outcome: Change in Reported Subjective Benefit on the Speech Domain of the Speech, Spatial and Qualities of Hearing (SSQ) Scale Over Time
Description: Participants reported subjective device benefit when hearing speech in a variety of competing contexts by marking on a visual analog scale from 0 to 10, with 0 being the minimum benefit and 10 being maximal benefit. Participants based their report on daily listening with the cochlear implant on and contralateral ear open. A higher score is greater subjective benefit reported by the participant.
Time Frame: Intervals within the first 12 months of device use
Population: as for outcome 1
Measure: Mean (Full Range); unit: Scores on a scale
Arm/Group | Vestibular Schwannoma | Meniere's Disease
Number analyzed (Participants) | 5 | 3
Scores on a scale
  1-Month | 6.2 [4 to 8.3] | 6.1 [4 to 7.8]
  3-Month | 6.6 [5.2 to 7.8] | 5.8 [3.6 to 8.4]
  6-Month | 6.8 [5.2 to 8.5] | 7.1 [6.1 to 8.4]
  12-Month: number analyzed (Participants) | 5 | 2
  12-Month | 5.4 [3.1 to 7.1] | 7.5 [5.8 to 9.3]

11. Primary Outcome: Change in Reported Subjective Benefit on the Spatial Domain of the SSQ Scale Over Time
Description: Participants reported subjective device benefit for the directional, distance, and movement components of spatial hearing by marking on a visual analog scale from 0 to 10, with 0 being the minimum benefit and 10 being maximal benefit. Participants based their report on daily listening with the cochlear implant on and contralateral ear open. A higher score is greater subjective benefit reported by the participant.
Time Frame: Intervals within the first 12 months of device use
Population: as for outcome 1
Measure: Mean (Full Range); unit: Score on a scale
Arm/Group | Vestibular Schwannoma | Meniere's Disease
Number analyzed (Participants) | 5 | 3
Score on a scale
  1-Month | 5.4 [2.5 to 6.9] | 6.4 [6 to 6.9]
  3-Month | 6 [4.9 to 6.8] | 7.5 [6.4 to 8.5]
  6-Month | 5.6 [3.9 to 6.6] | 7 [6.1 to 8.9]
  12-Month: number analyzed (Participants) | 5 | 2
  12-Month | 5.4 [3.1 to 7.1] | 7.5 [5.8 to 9.3]

12. Primary Outcome: Change in Reported Subjective Benefit on the Qualities of Hearing Domain of the SSQ Scale Over Time
Description: Participants reported subjective device benefit in qualities of hearing (including ease of listening and the naturalness, clarity, and identifiability of different sounds) by marking on a visual analog scale from 0 to 10, with 0 being the minimum benefit and 10 being maximal benefit. Participants based their report on daily listening with the cochlear implant on and contralateral ear open. A higher score is greater subjective benefit reported by the participant.
Time Frame: Intervals within the first 12 months of device use
Population: as for outcome 1
Measure: Mean (Full Range); unit: Score on a scale
Arm/Group | Vestibular Schwannoma | Meniere's Disease
Number analyzed (Participants) | 5 | 3
Score on a scale
  1-Month | 6.4 [3 to 10] | 5 [3 to 7]
  3-Month | 7.9 [6.6 to 9.6] | 7.2 [6.4 to 8.6]
  6-Month | 6.4 [1.6 to 9.9] | 7.3 [6.4 to 8.7]
  12-Month: number analyzed (Participants) | 5 | 2
  12-Month | 5.4 [3.1 to 7.1] | 7.5 [5.8 to 9.3]

13. Primary Outcome: Change in Reported Subjective Difficulty Frequency on the Abbreviated Profile of Hearing Aid Benefit (APHAB) Over Time
Description: Participants reported frequency of subjective difficulty in specific listening situations. Participants based their report on daily listening with the cochlear implant on and contralateral ear open. The score is percentage of how frequently participants experience difficulty in specific listening situations, ranging from 1% (Never) to 99% (Always). A lower global score is less reported difficulty frequency by the participant.
Time Frame: Intervals within the first 12 months of device use
Population: as for outcome 1
Measure: Mean (Full Range); unit: Percentage of situations with difficulty
Arm/Group | Vestibular Schwannoma | Meniere's Disease
Number analyzed (Participants) | 5 | 3
Percentage of situations with difficulty
  1-Month | 23.3 [9.7 to 38.7] | 37.8 [18.5 to 66.4]
  3-Month | 23.3 [11 to 39.3] | 25.4 [12.8 to 45.8]
  6-Month | 27.8 [5.9 to 59.4] | 24.6 [13.7 to 31.8]
  12-Month: number analyzed (Participants) | 5 | 2
  12-Month | 20.1 [6.5 to 35.1] | 16 [14.3 to 17.7]

14. Secondary Outcome: Difference in AzBio Sentences in Quiet Scores With the Cochlear Implant on (Plus Contralateral Ear Open) Versus Off (Contralateral Ear Alone) Over Time
Description: Testing open-set sentence understanding with no background noise present. Recorded AzBio Sentences lists were presented to the participant while listening with the cochlear implant on and contralateral ear open and also while listening with the cochlear implant off/contralateral ear alone; the speech and noise were collocated in this condition. Resultant score is a difference in mean percentage of words correct between cochlear implant on versus off; a positive difference translates to a higher score with the cochlear implant on, whereas a negative difference translates to a lower score with the cochlear implant on.
Time Frame: Intervals within the first 12 months of device use
Population: as for outcome 1
Measure: Mean (Full Range); unit: Percentage correct words
Arm/Group | Vestibular Schwannoma | Meniere's Disease
Number analyzed (Participants) | 5 | 3
Percentage correct words
  1-Month | 1 [-2 to 4] | 2.3 [0 to 6]
  3-Month | 0 [-1 to 1] | 0 [-1 to 1]
  6-Month | 0.2 [-3 to 5] | 0.7 [0 to 2]
  12-Month: number analyzed (Participants) | 5 | 2
  12-Month | 0.6 [0 to 3] | 0.5 [0 to 1]

15. Secondary Outcome: Difference in AzBio Sentences in Noise Scores (S0N0) With the Cochlear Implant on (Plus Contralateral Ear Open) Versus Off (Contralateral Ear Alone) Over Time
Description: Testing open-set sentence understanding with concurrent background noise present at 0 dB SNR. Recorded AzBio Sentences lists were presented to the participant while listening with the cochlear implant on and contralateral ear open and also while listening with the cochlear implant off/contralateral ear alone; the speech and noise were colocated in this condition (S0N0). Resultant score is a difference in the mean percentage of words correct between cochlear implant on versus off; a positive score translates to a higher score with the cochlear implant on, whereas a negative difference translates to a lower difference with the cochlear implant on.
Time Frame: Intervals within the first 12 months of device use
Population: as for outcome 1
Measure: Mean (Full Range); unit: Percentage correct words
Arm/Group | Vestibular Schwannoma | Meniere's Disease
Number analyzed (Participants) | 5 | 3
Percentage correct words
  1-Month | -3.6 [-14 to 15] | 1 [0 to 3]
  3-Month | -2.6 [-14 to 13] | -7.7 [-17 to 7]
  6-Month | -6.4 [-35 to 12] | -6 [-14 to 4]
  12-Month: number analyzed (Participants) | 5 | 2
  12-Month | -0.4 [-7 to 9] | 6 [-8 to 20]

16. Secondary Outcome: Difference in AzBio Sentences in Noise Scores (S0NCI) With the Cochlear Implant on (Plus Contralateral Ear Open) Versus Off (Contralateral Ear Alone) Over Time
Description: Testing open-set sentence understanding with concurrent background noise present at 0 dB SNR. Recorded AzBio Sentences lists were presented to the participant while listening with the cochlear implant on and contralateral ear open and also while listening with the cochlear implant off/contralateral ear alone; the speech was presented at 0 degrees azimuth and noise to the implanted side in this condition (S0NCI). Resultant score is a difference in mean percentage of words correct between cochlear implant on versus off; a positive difference translates to a higher score with the cochlear implant on, whereas a negative difference translates to a lower score with the cochlear implant on.
Time Frame: Intervals within the first 12 months of device use
Population: as for outcome 1
Measure: Mean (Full Range); unit: Percentage correct words
Arm/Group | Vestibular Schwannoma | Meniere's Disease
Number analyzed (Participants) | 5 | 3
Percentage correct words
  1-Month | 1.6 [-9 to 12] | -1.3 [-10 to 5]
  3-Month | -10.2 [-19 to -1] | 4.7 [1 to 9]
  6-Month | 4.4 [-9 to 27] | -4 [-8 to 0]
  12-Month: number analyzed (Participants) | 5 | 2
  12-Month | 0.8 [-7 to 7] | -2 [-9 to 5]

17. Secondary Outcome: Difference in AzBio Sentences in Noise Scores (S0NContra) With the Cochlear Implant on (Plus Contralateral Ear Open) Versus Off (Contralateral Ear Alone) Over Time
Description: Testing open-set sentence understanding with concurrent background noise present at 0 dB SNR. Recorded AzBio Sentences lists were presented to the participant while listening with the cochlear implant on and contralateral ear open and also while listening with the cochlear implant off/contralateral ear alone; the speech was presented at 0 degrees azimuth and noise to the contralateral ear in this condition (S0NContra). Resultant score is a difference in mean percentage of words correct between cochlear implant on versus off; a positive difference translates to a higher score with the cochlear implant on, whereas a negative difference translates to a lower score with the cochlear implant on.
Time Frame: Intervals within the first 12 months of device use
Population: as for outcome 1
Measure: Mean (Full Range); unit: Percentage correct words
Arm/Group | Vestibular Schwannoma | Meniere's Disease
Number analyzed (Participants) | 5 | 3
Percentage correct words
  1-Month | 10 [0 to 18] | -2.3 [-29 to 13]
  3-Month | 5.2 [-7 to 13] | 14.7 [8 to 25]
  6-Month | 9.6 [2 to 20] | 12.3 [11 to 14]
  12-Month: number analyzed (Participants) | 5 | 2
  12-Month | 10.4 [6 to 17] | 24.5 [19 to 30]

18. Secondary Outcome: Difference in BKB-SIN Scores (S0N0) With the Cochlear Implant on (Plus Contralateral Ear Open) Versus Off (Contralateral Ear Alone) Over Time
Description: Testing open-set sentence understanding with concurrent background noise present at various levels. Recorded BKB-SIN lists were presented to the participant while listening with the cochlear implant on and contralateral ear open and also while listening with the cochlear implant off/contralateral ear alone; the speech and noise were colocated in this condition (S0N0). Resultant score is a difference in the mean signal-to-noise ratio at which the participant scores 50% of the target words correct between cochlear implant on versus off; a negative difference translates to a better score with the cochlear implant on, whereas a positive difference translates to a worse score with the cochlear implant on.
Time Frame: Intervals within the first 12 months of device use
Population: as for outcome 1
Measure: Mean (Full Range); unit: dB SNR
Arm/Group | Vestibular Schwannoma | Meniere's Disease
Number analyzed (Participants) | 5 | 3
dB SNR
  1-Month | -1.5 [-4 to 1] | -0.3 [-1.5 to 0.5]
  3-Month | -0.8 [-3 to 1] | 1 [1 to 1]
  6-Month | 0.3 [-1.5 to 2] | -0.8 [-1.5 to 0.5]
  12-Month: number analyzed (Participants) | 5 | 2
  12-Month | -0.6 [-2 to 0] | -1 [-2 to 0]

19. Secondary Outcome: Difference in BKB-SIN Scores (S0NCI) With the Cochlear Implant on (Plus Contralateral Ear Open) Versus Off (Contralateral Ear Alone) Over Time
Description: Testing open-set sentence understanding with concurrent background noise present at various levels. Recorded BKB-SIN lists were presented to the participant while listening with the cochlear implant on and contralateral ear open and also while listening with the cochlear implant off/contralateral ear alone; the speech was presented at 0 degrees azimuth and noise to the implanted side in this condition (S0NCI). Resultant score is a difference in the mean signal-to-noise ratio at which the participant scores 50% of the target words correct between cochlear implant on versus off; a negative difference translates to a better score with the cochlear implant on, whereas a positive difference translates to a worse score with the cochlear implant on.
Time Frame: Intervals within the first 12 months of device use
Population: as for outcome 1
Measure: Mean (Full Range); unit: dB SNR
Arm/Group | Vestibular Schwannoma | Meniere's Disease
Number analyzed (Participants) | 5 | 3
dB SNR
  1-Month | 1.4 [0.5 to 2.5] | -0.5 [-1 to 0]
  3-Month | 0.4 [-1 to 3] | -0.2 [-1 to 1.5]
  6-Month | -0.6 [-3 to 1] | 0.5 [0 to 1]
  12-Month: number analyzed (Participants) | 5 | 2
  12-Month | -1.2 [-3 to 0] | -1.8 [-6 to 2.5]

20. Secondary Outcome: Difference in BKB-SIN Scores (S0NContra) With the Cochlear Implant on (Plus Contralateral Ear Open) Versus Off (Contralateral Ear Alone) Over Time
Description: Testing open-set sentence understanding with concurrent background noise present at various levels. Recorded BKB-SIN lists were presented to the participant while listening with the cochlear implant on and contralateral ear open and also while listening with the cochlear implant off/contralateral ear alone; the speech was presented at 0 degrees azimuth and noise to the contralateral ear in this condition (S0NContra). Resultant score is a difference in the mean signal-to-noise ratio at which the participant scores 50% of the target words correct between cochlear implant on versus off; a negative difference translates to a better score with the cochlear implant on, whereas a positive difference translates to a worse score with the cochlear implant on.
Time Frame: Intervals within the first 12 months of device use
Population: as for outcome 1
Measure: Mean (Full Range); unit: dB SNR
Arm/Group | Vestibular Schwannoma | Meniere's Disease
Number analyzed (Participants) | 5 | 3
dB SNR
  1-Month | 0.8 [-0.5 to 3] | -1.5 [-2.5 to 0]
  3-Month | -0.4 [-2 to 0.5] | -3 [-4 to -2.5]
  6-Month | -0.3 [-1 to 1.5] | -1.2 [-2.5 to 1.5]
  12-Month: number analyzed (Participants) | 5 | 2
  12-Month | -0.5 [-2 to 1] | 0.3 [0 to 0.5]

21. Secondary Outcome: Difference in Localization RMS Error With the Cochlear Implant on (Plus Contralateral Ear Open) Versus Off (Contralateral Ear Alone) Over Time
Description: Participants identified a speech-shaped noise source presented at various presentation levels within an 11-speaker array. Participants localized the sound source with the cochlear implant on and contralateral ear open and also while listening with the cochlear implant off/contralateral ear alone. The RMS error (degrees) was estimated; a lower degree is more accurate/better localization of the sound source. The resultant score reported here is a difference in mean RMS error between cochlear implant on versus off; a negative difference translates to a better score with the cochlear implant on, whereas a positive difference translates to a worse score with the cochlear implant on.
Time Frame: Intervals within the first 12 months of device use
Population: as for outcome 1
Measure: Mean (Full Range); unit: Degrees
Arm/Group | Vestibular Schwannoma | Meniere's Disease
Number analyzed (Participants) | 5 | 3
Degrees
  1-Month | -37.5 [-62.4 to -17.3] | -26.8 [-30.2 to -24.1]
  3-Month | -31.2 [-53.2 to -8.4] | -41.3 [-61 to -31.3]
  6-Month | -35.9 [-60.3 to -3.5] | -41.5 [-57.3 to -30.4]
  12-Month: number analyzed (Participants) | 5 | 2
  12-Month | -40 [-62.9 to -18.4] | -36.5 [-41.2 to -31.7]

ADVERSE EVENTS:
Time Frame: Data were collected from the time a participant was enrolled until the study endpoint, 12-months post-initial activation. Approximately 13 months in total for each participant.
Description: Adverse events were those events described as potential risks of the protocol. Serious adverse events were those events associated with the device that related to the rights, safety or welfare of participants.
Arm/Group | Vestibular Schwannoma | Meniere's Disease
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/3
Serious Adverse Events (participants affected / at risk) | 2/7 | 0/3
Other Adverse Events (participants affected / at risk) | 4/7 | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vestibular Schwannoma (N=7) | Meniere's Disease (N=3)
Unsuccessful Initial Activation (Ear and labyrinth disorders) | 2 | 0 — Participant denied auditory percept on all electrodes during initial activation of the study device.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vestibular Schwannoma (N=7) | Meniere's Disease (N=3)
Facial nerve weakness (Nervous system disorders) | 3 | 0 — Participants reported facial weakness on the implanted side.
Metallic taste on tongue on implanted side (Nervous system disorders) | 1 | 0 — Participants reported a metallic taste on their tongue on the side of the implant following surgery.
Fever and congestion (General disorders) | 0 | 1 — Participant reported onset of fever and congestion during cochlear implant device use.
"Unsettling feelings" reported (Psychiatric disorders) | 0 | 1 — Participant reported "unsettling feelings"; specifically, participant reported having a hard time concentrating and thinking clearly. Participant reported a history of depression before enrollment.
Nasal drainage and itching in noise (Immune system disorders) | 0 | 1 — Participant reported bilateral nasal drainage and sneezing/itching nostrils; participant reported a history of allergies prior to enrollment.
Migration of receiver/stimulator portion of cochlear implant (Product Issues) | 1 | 0 — Participant reported the cochlear implant's receiver/stimulator migrating.
Dizziness (Ear and labyrinth disorders) | 1 | 0 — Participant reported constant dizziness following surgery; participant previously reported a history of dizziness prior to enrollment.
Aural pressure (Ear and labyrinth disorders) | 1 | 0 — Participant reported feeling aural pressure around the external portion of the ear that was implanted following surgery.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-05-25): https://cdn.clinicaltrials.gov/large-docs/99/NCT02309099/Prot_SAP_000.pdf